CLINICAL TRIAL: NCT02778399
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2b Dose-ranging Study to Assess the Efficacy and Safety of OBE2109 in Subjects With Endometriosis Associated Pain
Brief Title: A Study to Assess the Efficacy and Safety of OBE2109 in Subjects With Endometriosis
Acronym: EDELWEISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-OBE2109-001
Record Dates: First submitted 2016-05-03; First posted 2016-05-19 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Endometriosis
Keywords: Pelvic Pain; Endometriosis; Dysmenorrhea; Dyspareunia
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea; Dyspareunia | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- OBE2109 50 mg (Experimental)
  Interventions: Drug: OBE2109
- OBE2109 75mg fixed dose (FD) (Experimental)
  Interventions: Drug: OBE2109
- OBE2109 75mg titrated dose (TD) (Experimental)
  Interventions: Drug: OBE2109
- OBE2109 100mg (Experimental)
  Interventions: Drug: OBE2109
- OBE2109 200 mg (Experimental)
  Interventions: Drug: OBE2109
- Placebo / OBE2109 100mg (Placebo Comparator): Participants received placebo for the first 12 weeks and were then crossed-over to active treatment with OBE2109 100mg for a further 12 weeks.
  Interventions: Drug: Placebo; Drug: OBE2109

INTERVENTIONS:
Drug: Placebo — Placebo tablets for oral administration once daily
  Arms: Placebo / OBE2109 100mg
Drug: OBE2109 — OBE2109 tablets for oral administration once daily

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of a range of oral doses of OBE2109 versus placebo, in reducing endometriosis associated pain.

DETAILED DESCRIPTION:
The study is a prospective, dose-finding, randomized, parallel group, double-blind, placebo-controlled phase 2b study investigating the efficacy and safety of OBE2109 in the treatment of 330 women with moderate-to-severe endometriosis associated pain.

Subject will be randomized to one of 6 treatment groups in a 1:1:1:1:1:1 ratio (1 placebo group, 5 dose groups with different dosage/regimen).

Eligible subjects will be offered the opportunity to continue treatment with OBE2109 in an extension phase. Subjects who do not continue in the extension will enter the treatment-free follow-up phase of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject must have had her most recent surgical and - if available - histological, diagnosis of pelvic endometriosis up to 10 years before screening.
* The subject has moderate to severe endometriosis-associated pain during the screening period.
* The subject has regular menstrual cycles.
* The subject has a BMI ≥ 18 kg/m2 at the screening visit.

Key Exclusion Criteria:

* The subject is pregnant or breast feeding or is planning a pregnancy within the duration of the treatment period of the study.
* The subject had an interventional surgery for endometriosis performed within a period of 60 days before screening.
* The subject did not respond to prior treatment with gonadotropin releasing hormone (GnRH) agonists or GnRH antagonists for endometriosis.
* The subject has a history of, or known osteoporosis or other metabolic bone disease.
* The subject has chronic pelvic pain that is not caused by endometriosis and requires chronic analgesic / therapy, or that would interfere with the assessment of endometriosis related pain.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (86):
- United States (71):
  - Site reference ID 455, Chandler, Arizona
  - Site reference ID 439, Scottsdale, Arizona
  - Site reference ID 462, Arcadia, California
  - Site reference ID 405, Chino, California
  - Site reference ID 463, Huntington Park, California
  - Site refenrec ID 469, Northridge, California
  - Site reference ID 431, San Diego, California
  - Site reference ID 440, Tustin, California
  - Site reference ID 474, Denver, Colorado
  - Site reference ID 450, Lakewood, Colorado
  - Site reference ID 425, Longmont, Colorado
  - Site reference ID 410, Washington D.C., District of Columbia
  - Site reference ID 457, Boca Raton, Florida
  - Site reference ID 418, Clearwater, Florida
  - Site reference ID 437, Gainesville, Florida
  - Site reference ID 458, Jensen Beach, Florida
  - Site reference ID 411, Miami, Florida
  - Site reference ID 424, Miami, Florida
  - Site reference ID 435, Miami, Florida
  - Site reference ID 420, Miami Lakes, Florida
  - Site reference ID 441, Miami Springs, Florida
  - Site reference ID 423, New Port Richey, Florida
  - Site reference ID 426, Tampa, Florida
  - Site reference ID 442, Wellington, Florida
  - Site reference ID 428, Atlanta, Georgia
  - Site reference ID 459, Atlanta, Georgia
  - Site reference ID 475, Nampa, Idaho
  - Site reference ID 465, Oak Brook, Illinois
  - Site reference ID 404, Shawnee Mission, Kansas
  - Site reference ID 456, Wichita, Kansas
  - Site reference ID 454, Marrero, Louisiana
  - Site reference ID 453, Metairie, Louisiana
  - Site reference ID 478, Glen Burnie, Maryland
  - Site reference ID 445, Fall River, Massachusetts
  - Site reference ID 471, Fall River, Massachusetts
  - Site reference ID 430, Ann Arbor, Michigan
  - Site reference ID 409, Bay City, Michigan
  - Site reference ID 468, Saginaw, Michigan
  - Site reference ID 473, Saginaw, Michigan
  - Site reference ID 427, Southfield, Michigan
  - Site reference ID 421, Albuquerque, New Mexico
  - Site reference ID 466, New York, New York
  - Site reference ID 436, Greensboro, North Carolina
  - Site reference ID 433, Morehead City, North Carolina
  - Site reference ID 443, Dayton, Ohio
  - Site reference ID 472, Franklin, Ohio
  - Site reference ID 415, Tiffin, Ohio
  - Site reference ID 414, Westerville, Ohio
  - Site reference ID 419, Bryn Mawr, Pennsylvania
  - Site reference ID 449, Jenkintown, Pennsylvania
  - Site reference ID 476, Columbia, South Carolina
  - Site reference ID 408, Bristol, Tennessee
  - Site reference ID 403, Chattanooga, Tennessee
  - Site reference ID 429, Nashville, Tennessee
  - Site reference ID 452, Austin, Texas
  - Site reference ID 461, Beaumont, Texas
  - Site reference ID 447, Dallas, Texas
  - Site reference ID 460, Dallas, Texas
  - Site reference ID 464, Fort Worth, Texas
  - Site reference ID 413, Houston, Texas
  - Site reference ID 434, Houston, Texas
  - Site reference ID 479, Houston, Texas
  - Site reference ID 451, San Antonio, Texas
  - Site reference ID 402, Schertz, Texas
  - Site reference ID 432, Webster, Texas
  - Site reference ID 422, Draper, Utah
  - Site reference ID 467, Centreville, Virginia
  - Site reference ID 407, Norfolk, Virginia
  - Site reference ID 412, Richmond, Virginia
  - Site reference ID 417, Richmond, Virginia
  - Site reference ID 406, Seattle, Washington
- Poland (5):
  - Site reference ID 101, Katowice
  - Site reference ID 102, Katowice
  - Site reference ID 104, Lublin
  - Site reference ID 105, Lublin
  - Site reference ID 103, Szczecin
- Russia (5):
  - Site reference ID 201, Moscow
  - Site reference ID 202, Moscow
  - Site reference ID 203, Moscow
  - Site reference ID 204, Moscow
  - Site reference ID 205, Saint Petersburg
- Ukraine (5):
  - Site reference ID 305, Ivano-Frankivsk
  - Site reefrence ID 303, Kyiv
  - Site reference ID 301, Kyiv
  - Site reference ID 302, Kyiv
  - SIte reference ID 304, Kyiv

REFERENCES:
- [Derived] Donnez J, Taylor HS, Taylor RN, Akin MD, Tatarchuk TF, Wilk K, Gotteland JP, Lecomte V, Bestel E. Treatment of endometriosis-associated pain with linzagolix, an oral gonadotropin-releasing hormone-antagonist: a randomized clinical trial. Fertil Steril. 2020 Jul;114(1):44-55. doi: 10.1016/j.fertnstert.2020.02.114. Epub 2020 Jun 4. PMID 32505383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 328 females were randomized at 62 sites in 4 countries: 48 sites in USA (177 subjects), 5 sites in Poland (67 subjects), 5 sites in Ukraine (73 subjects) and 4 sites in Russia (11 subjects).
Pre-assignment Details: 716 subjects were screened and 328 were randomized; 327 were included in the safety set (1 not included as didn't receive study treatment). 323 subjects were included in the Full Analysis Set (FAS), 5 randomized subjects were excluded: 1 as per the safety set and 4 were prematurely discontinued at one US site due to the site's serious non-compliance to the protocol.
Groups:
- Placebo / OBE2109 100mg: Placebo: Placebo tablets for oral administration once daily.
  OBE2109: OBE2109 tablets for oral administration once daily. Participants received placebo for the first 12 weeks and were then crossed-over to active treatment with OBE2109 100mg for a further 12 weeks.
- OBE2109 50mg; OBE2109 100mg; OBE2109 200mg: OBE2109 tablets for oral administration once daily
- OBE2109 75mg FD: OBE2109 tablets for oral administration once daily. FD = Fixed Dose
- OBE2109 75mg TD: OBE2109 tablets for oral administration once daily. TD = Titrated Dose
Period: Up to Week 12 Treatment Period
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Started | 54 | 49 | 57 | 58 | 53 | 57
Included in SAFETY SET | 54 | 49 | 57 | 58 | 52 | 57
Included in FAS | 53 | 49 | 56 | 58 | 51 | 56
Completed | 45 | 45 | 53 | 51 | 45 | 49
Not Completed | 9 | 4 | 4 | 7 | 8 | 8
Not completed — Adverse Event | 1 | 2 | 3 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 5 | 2 | 1 | 4 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0 | 2
Not completed — other - reason not stated | 0 | 0 | 0 | 1 | 2 | 0
Period: Week 12 to Week 24 Treatment Period
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Started | 45 | 45 | 53 | 51 | 45 | 49
Completed | 37 | 41 | 48 | 46 | 39 | 42
Not Completed | 8 | 4 | 5 | 5 | 6 | 7
Not completed — Adverse Event | 2 | 0 | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 3 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 1 | 0 | 2 | 0 | 0 | 0
Not completed — other - reason not stated | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- OBE2109 75mg FD; OBE2109 75mg TD; OBE2109 100mg; OBE2109 200mg: OBE2109 tablets for oral administration once daily
- Total: Total of all reporting groups
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg | Total
Number analyzed (Participants) | 53 | 49 | 56 | 58 | 51 | 56 | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 49 | 56 | 58 | 51 | 56 | 323
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.78) | 30.9 (5.98) | 32.0 (6.83) | 31.2 (5.85) | 33.0 (5.78) | 30.9 (6.03) | 31.7 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 56 | 58 | 51 | 56 | 323
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 7 | 4 | 5 | 27
  Not Hispanic or Latino | 25 | 18 | 27 | 25 | 24 | 23 | 142
  Unknown or Not Reported | 25 | 26 | 26 | 26 | 23 | 28 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 5 | 8 | 3 | 3 | 25
  White | 49 | 46 | 50 | 50 | 46 | 52 | 293
  More than one race | 0 | 1 | 1 | 0 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 30% or Greater Reduction From Baseline to Week 12 in Mean Overall Pelvic Pain Score (0-3 VRS)
Description: The primary efficacy endpoint of the study was a response at Week 12, with response defined as a reduction of 30% or greater from baseline in the mean overall pelvic pain score, defined as the mean of daily pain scores reported in electronic diary during the preceding 28 days (4-week period), assessed on a Verbal Rating Scale for pelvic pain of 0 (no pain) to 3 (severe pain). The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: Number of subjects with available score in the respective group, from the Full Analysis Set (All randomized subjects who received at least one dose of study drug and had at least one assessment after first dose).
  Data for the 75mg group (FD) and 75mg titrated group (TD) were combined for the analyses of the first 12 weeks of treatment, as pre-specified in the protocol (section 9.5).
Measure: Number; unit: percentage of subjects
Groups:
- OBE2109 75mg FD + TD; OBE2109 100mg; OBE2109 200mg: OBE2109 tablets for oral administration once daily
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
percentage of subjects | 34.5 | 49.4 | 61.5 | 56.4 | 56.3

2. Secondary Outcome: Change From Baseline to Week 12 in the Mean Overall Pelvic Pain Score (0-10 NRS)
Description: This endpoint corresponds to the change from baseline to Week 12 in the mean overall pelvic pain score, defined as the mean of daily pain scores reported in electronic diary during the preceding 28 days (4-week period), assessed on a Numerical Rating Scale (NRS) for pelvic pain of 0 (no pelvic pain) to 10 (worst pelvic pain imaginable). The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
score on a scale | -1.17 [-1.70 to -0.65] | -1.75 [-2.29 to -1.20] | -2.15 [-2.50 to -1.80] | -2.06 [-2.60 to -1.52] | -2.14 [-2.65 to -1.63]

3. Secondary Outcome: Percentage of Subjects With 30% or Greater Reduction From Baseline to Week 12 in Mean Pelvic Pain Scores (0-3 VRS) for Days With Uterine Bleeding
Description: This endpoint corresponds to a response at Week 12, with response defined as a reduction of 30% or greater from baseline in the mean pelvic pain score for days with uterine bleeding/spotting, defined as the mean of daily pain scores on days with uterine bleeding/spotting recorded in electronic diary during the preceding 28 days (4-week period), assessed on a Verbal Rating Scale for pelvic pain of 0 (no pain) to 3 (severe pain). The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
percentage of subjects | 28.5 | 43.3 | 68.2 | 68.6 | 78.9

4. Secondary Outcome: Percentage of Subjects With 30% or Greater Reduction From Baseline to Week 12 in Mean Pelvic Pain Scores (0-3 VRS) for Days With no Uterine Bleeding
Description: This endpoint corresponds to a response at Week 12, with response defined as a reduction of 30% or greater from baseline in the mean pelvic pain score for days with no uterine bleeding, defined as the mean of daily pain scores on days with no uterine bleeding recorded in electronic diary during the preceding 28 days (4-week period) on a Verbal Rating Scale for pelvic pain of 0 (no pain) to 3 (severe pain). The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 50 | 55
percentage of subjects | 37.1 | 46.2 | 58.5 | 61.5 | 47.7

5. Secondary Outcome: Change From Baseline to Week 12 in the Mean Dyspareunia Score (0-3 VRS)
Description: This endpoint corresponds to the change from baseline to Week 12 in the mean dyspareunia score, defined as the mean of daily dyspareunia scores recorded in electronic diary during the preceding 28 days (4-week period), assessed on a 0-3 Verbal Rating Scale (VRS) for dyspareunia, with 0 representing "No discomfort during sexual intercourse" and 3 representing "I avoided sexual intercourse because of pain". The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The dyspareunia questionnaire also included an option "not applicable: I was not sexually active for reasons other than my endometriosis or did not have sexual intercourse"; for scoring, answering "not applicable" was considered like a missing value.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 47 | 40 | 90 | 44 | 44
score on a scale | -0.39 [-0.63 to -0.16] | -0.62 [-0.87 to -0.37] | -0.59 [-0.76 to -0.43] | -0.66 [-0.91 to -0.41] | -0.79 [-1.03 to -0.54]

6. Secondary Outcome: Change From Baseline to Week 12 in the Mean Dyschezia Score (0-10 NRS)
Description: This endpoint corresponds to the change from baseline to week 12 in the mean dyschezia score, defined as the mean of weekly dyschezia scores reported in electronic diary during the preceding 28 days (4-week period), assessed on a 0-10 Numerical Rating Scale for dyschezia, with 0 representing no pain and 10 representing the worst pain imaginable. The baseline mean score was calculated as the mean of weekly scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale/week
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 113 | 50 | 55
score on a scale/week | -0.78 [-1.34 to -0.22] | -1.55 [-2.14 to -0.96] | -1.87 [-2.25 to -1.49] | -1.97 [-2.55 to -1.39] | -1.7 [-2.25 to -1.15]

7. Secondary Outcome: Percentage of Subjects With Any Analgesics Use at Week 12
Description: This endpoint corresponds to the percentage of subjects at week 12 who recorded at least one pain medication intake in electronic diary during the preceding 28 days (4-week period).
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Placebo / OBE2109 100mg: Placebo: Placebo tablets for oral administration once daily
  OBE2109: OBE2109 tablets for oral administration once daily. Participants received placebo for the first 12 weeks and were then crossed-over to active treatment with OBE2109 100mg for a further 12 weeks
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
percentage of subjects | 90.6 [78.6 to 96.2] | 77.1 [62.7 to 87.1] | 74.8 [65.7 to 82.1] | 68.8 [54.1 to 80.5] | 72.1 [58.4 to 82.7]

8. Secondary Outcome: Change From Baseline to Week 12 in the Mean Score of Endometriosis Health Profile-30 (EHP-30) Pain Domain
Description: This endpoint corresponds to the change from baseline to Week 12 in the mean score of pain dimension of the EHP-30. The EHP-30 questionnaire was answered on electronic diary after activation by site staff during subject's monthly visits at site.
  The EHP-30 pain dimension consists of 11 items each addressing the effect of pain on various activities in the past 4 weeks and each assessed on a 5-point scale (0=Never through to 4=Always). Scaled score was equalled to total of raw score of each item in scale divided by the maximum possible raw score of all the items in the dimension, multiplied by 100, resulting in a score on a scale from 0 (best possible health status) to 100 (worst possible health status).
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 41 | 41 | 96 | 43 | 44
score on a scale | -7.4 [-12.36 to -2.41] | -18.5 [-23.44 to -13.47] | -18.9 [-22.20 to -15.69] | -19.4 [-24.28 to -14.55] | -20.9 [-25.69 to -16.10]

9. Secondary Outcome: Percentage of Subjects With Improvement in the Patient Global Impression of Change (PGIC) Score at Week 12
Description: The PGIC questionnaire consists of one question rated on a seven point scale (1="Very Much Improved" to 7="Very Much Worse"), with which the subject had to qualify her overall status since the start of the study. The PGIC was answered on electronic diary after activation by site staff during Week 12 visit at site.
  This endpoint corresponds to the percentage of subjects with an "improvement" in the PGIC score, which includes all subjects who answered "Very much improved" or "Much improved" or "Minimally improved" at Week 12.
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 43 | 42 | 98 | 43 | 46
percentage of subjects | 65.1 | 78.6 | 80.6 | 86 | 95.7

10. Secondary Outcome: Percentage of Subjects With an Endometriosis Severity Score of "Severe" at Week 12
Description: Subject was asked monthly on electronic diary to assess their impression of endometriosis severity, considering the preceding 4-weeks, with following possible answers: no symptoms, very mild, mild, moderate, severe. This question was programmed to raise automatically every 4 weeks on the subject electronic diary. Result reported here is the percentage of subjects who answered "severe" at week 12.
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
percentage of subjects | 20.9 | 4.5 | 7.8 | 4.5 | 4.2

11. Secondary Outcome: Change From Baseline to Week 12 in the Difficulty in Doing Daily Activities Mean Score
Description: This endpoint corresponds to the change from baseline to Week 12 in the mean of daily scores for "difficulty in doing daily activities", assessed via electronic diary during the preceding 28 days (4-week period), on a Numerical Rating Scale (NRS) of 0 (no difficulty doing daily activities) to 10 (unable to do daily activities). The baseline mean score was calculated as the mean of daily scores recorded in electronic diary over the two complete menstrual cycles performed during the screening period.
  The relevant time points are Baseline and Week 12.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD + TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 52 | 48 | 114 | 51 | 55
score on a scale | -1.17 [-1.68 to -0.65] | -1.65 [-2.18 to -1.12] | -2.06 [-2.41 to -1.72] | -1.88 [-2.41 to -1.36] | -1.99 [-2.49 to -1.49]

12. Secondary Outcome: Percentage Change From Baseline to Week 24 in Bone Mineral Density (BMD)
Description: Change from baseline to Week 24 in BMD assessed by dual-energy X-ray absorptiometry (DXA) scan of LUMBAR SPINE.
Time Frame: From baseline up to week 24
Population: Number of subjects with available BMD results at Week 24 in the respective group, from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 34 | 38 | 45 | 42 | 37 | 38
percentage change | -0.929 [-1.71 to -0.15] | 0.137 [-0.83 to 1.11] | -0.798 [-1.57 to -0.03] | -1.000 [-1.71 to -0.29] | -1.365 [-2.14 to -0.59] | -2.602 [-3.56 to -1.65]

13. Secondary Outcome: Number of Non Benign Endometrial Biopsies at Week 24
Description: Any pathological changes in the endometrium at week 24 were assessed from endometrial biopsies. The number of non benign biopsies at Week 24 is presented per treatment arm.
  Note: an isolated case of hyperplasia (without atypia) was observed at week 12 in the 200 mg group in a subject whose screening biopsy results were normal. A follow-up biopsy at week 24 revealed no abnormalities.
Time Frame: Week 24
Population: Number of subjects with available endometrial biopsy result at Week 24 in the respective group (excluding those with tissue unsatisfactory for evaluation), from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Number; unit: Non benign biopsies
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 11 | 16 | 19 | 17 | 13 | 4
Non benign biopsies | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline to Week 24 in Endometrial Thickness Measured by Transvaginal Ultrasound (TVUS)
Description: The endometrium thickness was measured by TVUS at screening and at Week 24 visit by the gynaecologist and result was recorded in mm. This endpoint reports the changes from baseline to Week 24 in the endometrial thickness.
Time Frame: From baseline up to week 24
Population: Number of subjects with available TVUS result at Week 24 in the respective group, from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 35 | 41 | 49 | 45 | 39 | 41
mm | -3.1 (4.64) | -1.5 (4.28) | -2.3 (4.15) | -1.3 (3.70) | -1.6 (4.56) | -4.0 (3.39)

15. Secondary Outcome: Percentage Change From Baseline to Week 24 in the Clinical Laboratory Assessments: LDL
Description: This endpoint reports the change from baseline up to Week 24 in the clinical laboratory assessments: LDL cholesterol.
Time Frame: From baseline up to week 24
Population: Number of subjects with available laboratory LDL result at Week 24 in the respective group, from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 39 | 40 | 48 | 47 | 41 | 41
percent change | 1.7 (15.7) | -0.3 (16.6) | 7.4 (55.2) | 7.3 (21.4) | 9.7 (20.7) | 10.3 (21.7)

16. Secondary Outcome: Percentage Change From Baseline to Week 24 in Clinical Laboratory Assessments: HDL
Description: This endpoint reports the change from baseline to week 24 in clinical laboratory assessments: HDL cholesterol.
Time Frame: From Baseline up to week 24
Population: Number of subjects with available laboratory HDL result at Week 24 in the respective group, from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 39 | 40 | 48 | 47 | 41 | 41
percent change | 5.5 (11.7) | 2.9 (12.9) | 3.8 (17.8) | 6.2 (24.1) | 5.6 (18.0) | 8.1 (14.7)

17. Secondary Outcome: Percentage Change From Baseline to Week 24 in Clinical Laboratory Assessments: Triglycerides
Description: This endpoint reports the change from baseline to week 24 in clinical laboratory assessments: triglycerides.
Time Frame: From baseline up to week 24
Population: Number of subjects with available laboratory result for Triglycerides at Week 24 in the respective group, from the Safety Set (all randomized subjects who received at least one dose of double-blind study drug irrespective of the treatment received).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo / OBE2109 100mg | OBE2109 50mg | OBE2109 75mg FD | OBE2109 75mg TD | OBE2109 100mg | OBE2109 200mg
Number analyzed (Participants) | 39 | 40 | 48 | 47 | 41 | 41
percent change | 17.9 (38.6) | 16.4 (41.3) | 5.2 (35.2) | 13.6 (45.0) | 20.5 (80.6) | 24.0 (57.7)

ADVERSE EVENTS:
Time Frame: From baseline up to week 24
Groups:
- Placebo BL-Wk12: Placebo: Placebo tablets for oral administration once daily.
  In this arm, participants received placebo for the first 12 weeks, from baseline (BL) to week 12 (Wk12).
  They were then crossed-over to active treatment with OBE2109 100mg for a further 12 weeks (from week 12 to week 24, reported in separate group).
- OBE2109 100mg Wk12-Wk24: OBE2109: OBE2109 tablets for oral administration once daily.
  In this arm, participants received placebo for the first 12 weeks from baseline to week 12 (reported in separate group).
  They were then crossed-over to active treatment with OBE2109 100mg for a further 12 weeks, from week 12 (Wk12) to week 24 (Wk24).
- OBE2109 50mg BL-Wk24; OBE2109 75mg FD BL-Wk24; OBE2109 75mg TD BL-Wk24; OBE2109 100mg BL-Wk24; OBE2109 200mg BL-Wk24: OBE2109 tablets for oral administration once daily, from baseline (BL) to week 24 (Wk24)
Arm/Group | Placebo BL-Wk12 | OBE2109 100mg Wk12-Wk24 | OBE2109 50mg BL-Wk24 | OBE2109 75mg FD BL-Wk24 | OBE2109 75mg TD BL-Wk24 | OBE2109 100mg BL-Wk24 | OBE2109 200mg BL-Wk24
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/49 | 0/58 | 0/56 | 0/52 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/55 | 1/49 | 0/58 | 0/56 | 3/52 | 1/57
Other Adverse Events (participants affected / at risk) | 22/55 | 19/55 | 27/49 | 30/58 | 36/56 | 31/52 | 39/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BL-Wk12 (N=55) | OBE2109 100mg Wk12-Wk24 (N=55) | OBE2109 50mg BL-Wk24 (N=49) | OBE2109 75mg FD BL-Wk24 (N=58) | OBE2109 75mg TD BL-Wk24 (N=56) | OBE2109 100mg BL-Wk24 (N=52) | OBE2109 200mg BL-Wk24 (N=57)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BL-Wk12 (N=55) | OBE2109 100mg Wk12-Wk24 (N=55) | OBE2109 50mg BL-Wk24 (N=49) | OBE2109 75mg FD BL-Wk24 (N=58) | OBE2109 75mg TD BL-Wk24 (N=56) | OBE2109 100mg BL-Wk24 (N=52) | OBE2109 200mg BL-Wk24 (N=57)
abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 4 | 1
acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3 | 2 | 0 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 9
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 2 | 0 | 0
blood creatine phosphokinase increased (Investigations) | 1 | 1 | 1 | 4 | 5 | 2 | 4
bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 3
dizziness (Nervous system disorders) | 0 | 0 | 1 | 3 | 1 | 2 | 2
fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 2
headache (Nervous system disorders) | 14 | 9 | 12 | 10 | 16 | 15 | 17
hot flush (Vascular disorders) | 6 | 5 | 9 | 11 | 13 | 15 | 26
influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 3 | 0
libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3
mood swings (Psychiatric disorders) | 5 | 1 | 2 | 1 | 3 | 3 | 2
nasopharyngitis (Infections and infestations) | 3 | 1 | 8 | 7 | 4 | 2 | 1
nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | 2 | 4 | 7
pyrexia (General disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 3
toothache (Gastrointestinal disorders) | 3 | 1 | 3 | 2 | 0 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 3 | 2 | 5
vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
weight increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose study information which is not publicly available without prior written consent of Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02778399/Prot_SAP_000.pdf